CLINICAL TRIAL: NCT06312423
Title: Phase 1 Open-label Dose-escalation Study to Evaluate the Safety and Pharmacokinetics of IMT504 Phosphorothioate Oligonucleotide, an Immunomodulator and Tissue Repair Inducer, in Healthy Volunteers
Brief Title: Safety and Pharmacokinetics of IMT504, an Immunomodulator and Tissue Repair Inducer
Acronym: ECDA000/02
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ministry of Public Health of the Province of La Rioja (Other Government)
Collaborators: Immunalgia Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ECDA000/02
Record Dates: First submitted 2024-02-28; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Immune System
Keywords: INMUNOMODULATOR; OLIGONUCLEOTIDE; CYTOKINES
MeSH Terms: interventions — Phosphorothioate Oligonucleotides; IMT504

STUDY DESIGN:
Intervention Model Description: A total of 12 healthy adult volunteers of both sexes will be included, who will be progressively incorporated into 3 groups of 4 volunteers each. All volunteers will be evaluated at a research site authorized by the Regulatory Authority (ANMAT) to conduct phase 1 studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - 20 mg (Experimental): Four volunteers will be enrolled (no more than one per day and only after verifying that the preceding volunteer did not show any significant adverse effects) who will be administered the initial dose level (1 x 20 mg of IMT504).
  Interventions: Drug: Oligonucleotides, Phosphorothioate
- Group 2 - 60 mg (Experimental): If no toxicity is detected and there is good tolerance, another 4 patients will be enrolled (no more than one per day and only after verifying that the preceding one did not show significant adverse effects) who will receive treatment with the next dose level (3 x 20 mg of IMT504, one application per day for 3 consecutive days).
  Interventions: Drug: Oligonucleotides, Phosphorothioate
- Group 3 - 100 mg (Experimental): If no toxicity is detected and there is good tolerance, another 4 patients will be enrolled (no more than one per day and only after verifying that the preceding one did not show significant adverse effects) who will receive treatment with the next dose level (5 x 20 mg of IMT504, one application per day for 5 consecutive days).
  Interventions: Drug: Oligonucleotides, Phosphorothioate

INTERVENTIONS:
Drug: Oligonucleotides, Phosphorothioate — Group 1: 20 mg/day single dose Group 2: 20 mg/day for 3 days Group 3: 20 mg/day for 5 days
  Other Names: IMT504

SUMMARY:
Phase 1 open-label dose-escalation study to evaluate the safety and pharmacokinetics of IMT504 Phosphorothioate Oligonucleotide, an immunomodulator and tissue repair inducer, in healthy volunteers.

DETAILED DESCRIPTION:
This is a phase 1 open-label dose-escalation study to evaluate the safety and pharmacokinetics of IMT504 Phosphorothioate Oligonucleotide, an immunomodulator and tissue repair inducer, in healthy volunteers.

A total of 12 adult volunteers of both sexes will be included, who will be progressively incorporated into 3 groups of 4 volunteers each. The first group will be administered subcutaneously with a single dose of 20 mg of IMT504. The second group will receive 3 doses (20 mg daily for 3 days) and then, if no toxicity is detected, the last group will be administered 5 daily doses of 20 mg/d.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18 years or older.
2. With the capacity and willingness to comply with the prohibitions and restrictions specified in the protocol.
3. In female volunteers of childbearing potential, negative pregnancy test at the beginning of the study and commitment to using a contraceptive method from the date of consent signing until 3 months after the study is completed.
4. Capable of reading and understanding all the features of the study.
5. Negative PCR (Polymerase Chain reaction) for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2 ) virus;
6. Laboratory analysis without clinically significant variations within the 30 days prior to receiving the first dose of the investigational drug.
7. Negative serologies for hepatitis B virus (surface antigens [HBsAg] and antibodies against the core of hepatitis B virus [AntiHBc]), hepatitis C virus (AntiHCV), and human immunodeficiency virus (HIV).
8. Electrocardiogram (ECG) without evidence of acute or chronic significant pathologies.
9. Chest X-ray without significant pathological findings.
10. Capable of providing their signed and dated informed consent by the study volunteer and the authorized physician.

Exclusion Criteria:

1. Having participated in a research study within the 60 days prior to the start of the study.
2. Having a history of known allergies or a history of anaphylaxis or any other serious adverse reaction to any known drug or excipient.
3. History of alcoholism or substance abuse that would prevent compliance with the protocol characteristics.
4. Acute infectious disease at the time of enrollment or temperature ≥38.0°C in the 24 hours prior to the scheduled study vaccination.
5. Any laboratory abnormality with a severity grade >1 according to the Common Toxicity Criteria (CTC version 5 - November 2017).
6. Body Mass Index (BMI) greater than 35 kg/m2.
7. History of any active chronic disease.
8. Having received an investigational drug (including drugs related to COVID-19 prophylaxis or sepsis) or used an invasive investigational medical device in the 30 days prior to the start of the study.
9. Ongoing pregnancy or planned pregnancy within 3 months after administration of the investigational treatment, or lactation period.
10. Having undergone a surgical procedure requiring hospitalization in the 12 weeks prior to the start of the study, or not fully recovered from the surgery requiring hospitalization, or having a scheduled surgery requiring hospitalization during the expected study participation period or within 3 months after administration of the investigational treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety: Local and systemic reaction after administration of each dose of the investigational drug | Day 0, day 1 (group 1), days 1, 2, 3 (group 2) and days 1, 2, 3, 4, 5 (group 3), day 7 and day 28 after last administration of investigational drug
  Number of volunteers overall and in each dose group with local or systemic reaction, based on evaluation of adverse event recorded during clinical assessments
Safety: Serious adverse event | Day 0 to day 28 after last administration of investigational drug
  Number of volunteers overall and in each dose group with investigational drug - associated serious adverse events
Safety: Variations in the Laboratory results | Day 0, day 1 (group 1), days 1, 2, 3 (group 2) and days 1, 2, 3, 4, 5 (group 3) and day 7 after last administration of investigational drug
  Number of volunteers overall and in each dose group with variations in laboratory results from baseline to different control
Pharmacokinetics: IMT504 level in Serum | 0, 0.5, 1, 2, 4, 6, 8, 12, 24 hours after last administration of investigational drug
  Blood samples taken at different times to evaluate:
  - Maximum concentration (Cmax) defined as the maximum plasma concentration of the drug during a dosing interval (peak)
Pharmacokinetics: IMT504 level in Serum | 0, 0.5, 1, 2, 4, 6, 8, 12, 24 hours after last administration of investigational drug
  Blood samples taken at different times to evaluate:
  - Maximum time (tmax): time necessary to reach Cmax (Tmax).
Pharmacokinetics: IMT504 level in Serum | 0, 0.5, 1, 2, 4, 6, 8, 12, 24 hours after last administration of investigational drug
  Blood samples taken at different times to evaluate:
  - Area under the curve (AUC): defined as "total exposure", it is the area under the concentration-time curve, and represents a function of the total amount of bioavailable drug.
Pharmacokinetics: IMT504 level in Serum | 0, 0.5, 1, 2, 4, 6, 8, 12, 24 hours after last administration of investigational drug
  Blood samples taken at different times to evaluate:
  - Half time (t1/2): defined as the time to reduce the drug concentration by half.
Pharmacokinetics: IMT504 level in Serum | 0, 0.5, 1, 2, 4, 6, 8, 12, 24 hours after last administration of investigational drug
  Blood samples taken at different times to evaluate:
  - Clearance (CL): Plasma volume of the product that is cleared per unit of time.

SECONDARY OUTCOMES:
Pharmacodynamics: Interleukin - 35 | 0, 24 and 48 hours after last administration of investigational drug
  Blood samples taken at different point of evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Pirotzky, Doctor, Principal Investigator — Centro Nuestra Señora del Pilar; Alejandro Montaner, Doctor, Study Chair — Immunalgia Therapeutics S.A.
Locations (1):
- CENTRO DE INVESTIGACIÓN PARA ESTUDIOS DE FARMACOLOGÍA CLÍNICA DE FASE1 EN POBLACIÓN ADULTA y DE BIOEQUIVALENCIA. Sanatorio Nuestra Señora del Pilar, Buenos Aires, Argentina